CLINICAL TRIAL: NCT00662857
Title: A Phase 2, Open-Label, Randomized, 2-Way Crossover, Clinical Trial to Compare the Pharmacokinetics of 2 Formulations of "Intended Commercial Product" Technosphere® Insulin Inhalation Powder and to Determine the Bioavailability of a 30 Unit Cartridge of "Intended Commercial Product" Technosphere® Insulin Inhalation Powder Versus a 10 Unit Subcutaneous Injection of Insulin Lispro in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study Designed to Compare 2 Dose Strengths of TI Inhalation Powder in Adults With Type 1 Diabetes Mellitus and to Compare One of Those Formulations (30Units) With an Injection of Insulin Lispro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-116
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus: Type 1
Keywords: Diabetic adult male, diabetic adult female
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (3):
- 1: TI Inhalation Powder A (Experimental): Technosphere® Insulin Inhalation Powder, two 15 U cartridges
  Interventions: Drug: Technosphere® Insulin Inhalation Powder
- 2: TI Inhalation Powder B (Experimental): Technosphere® Insulin Inhalation Powder, one 30 U cartridge
  Interventions: Drug: Technosphere Insulin® Inhalation Powder
- 3: RAA Population (Experimental): Rapid Acting Analogue subjects received 10 IU sc Insulin Lispro
  Interventions: Drug: RAA Population

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation Powder — TI Inhalation Powder, two 15 U cartridges
  Arms: 1: TI Inhalation Powder A
Drug: Technosphere Insulin® Inhalation Powder — TI Inhalation Powder, one 30 U cartridge
  Arms: 2: TI Inhalation Powder B
Drug: RAA Population — RAA Population: All subjects received a single 10 IU sc injection of insulin lispro.
  Arms: 3: RAA Population

SUMMARY:
28 subjects to be enrolled for a screening period, 3 dosing visits & a follow-up visit. Visits 2 and 3 dosing of TI Inhalation Powder, cross over between two 15 U cartridges and one 30 U cartridge. Visit 4 dosing will be a sc injection of 10 IU of RAA (rapid-acting insulin analogue).

DETAILED DESCRIPTION:
28 eligible subjects were planned to be enrolled to determine bioequivalence and safety parameters of two 15 U TI Inhalation Powder cartridges versus one 30 U TI Inhalation Powder cartridge, according to a randomized, 2-way crossover design. Additionally, bioavailability of one 30 U TI Inhalation Powder cartridge to a single subcutaneous injection of 10 IU of RAA will be compared.

ELIGIBILITY:
Inclusion Criteria:

Males and Females > 18 and < 60 years of age Clinical diagnosis of type 1 diabetes mellitus with stable anti-diabetic regimen for at least 90 days prior to Screening BMI of < 30 kg/m2 Non-smokers (never smoked or former smokers (> 6 months since cessation) Pulmonary Function Testing (FEV1 > 70%, FEV1/FVC > 70%, TLC > 80% DLco [unc] > 70% of Predicted Written Informed consent

Exclusion Criteria:

Two or more severe hypoglycemic episodes within 6 months of Screening/Visit 1 Severe complications of diabetes Previous exposure to any inhaled insulin product other than TI inhalation Powder or similar formulation Inability to perform PFT maneuvers meeting recommended American Thoracic Society (ATS) standards of acceptability and repeatability criteria Respiratory tract infection within 8 weeks prior to Screening/Visit 1 History of chronic obstructive pulmonary disease (COPD), clinically proven asthma, and/or any other clinically important pulmonary disease (eg. Obstructive sleep apnea), confirmed by pulmonary function testing, and/or radiologic findings Major organ system diseases including seizures, heart failure, uncontrolled hypertension, cancer within the past 5 years, liver disease, anemia or autoimmune disorder Clinically significant abnormalities on screening laboratory evaluation Female subjects who are pregnant, lactating, or planning to become pregnant during the clinical trial period or not practicing adequate birth control Unable and/or unlikely to comprehend how to use the investigational device in this study or to follow study instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Profil Institute for Clinical Research Inc., Chula Vista, California
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single site with first subject screened 24 Apr 2008
Pre-assignment Details: Subjects assigned at Visit 2 to either: 2 15 U cartridges (TI Inhalation Powder A) or 1 30 U cartridge (TI Inhalation Powder B). At Visit 3 each subject was crossed over to the other treatment group. At Visit 4 subjects received a single sc injection of 10 IU of insulin lispro to 1 of 3 possible injection sites: arm, leg, or abdomen.
Groups:
- TI - A (2x15 U)/TI - B (1x30 U)/10 U sc Insulin Lispro: Treatment sequence: 30 U of Technosphere Insulin (TI) administered as 2 x 15 U cartridges as a single-dose, followed by 30 U of Technosphere Insulin (TI) administered as 1 x 30 U cartridges as a single-dose, and then 10 U of insulin lispro administered subcutaneously (sc) during a glucose clamp procedure
- TI - B (1x30 U)/TI - A (2x15 U)/10 U sc Insulin Lispro: Treatment sequence: 30 U of Technosphere Insulin (TI) administered as 1 x 30 U cartridges as a single-dose, followed by 30 U of Technosphere Insulin (TI) administered as 2 x 15 U cartridges as a single-dose, and then 10 U of insulin lispro administered subcutaneously (sc) during a glucose clamp procedure
Period: TI Dosing Period 1 (1 Day)
Arm/Group | TI - A (2x15 U)/TI - B (1x30 U)/10 U sc Insulin Lispro | TI - B (1x30 U)/TI - A (2x15 U)/10 U sc Insulin Lispro
Started | 13 | 16
Completed | 13 | 16
Not Completed | 0 | 0
Period: Washout 1 (3 - 14 Days)
Arm/Group | TI - A (2x15 U)/TI - B (1x30 U)/10 U sc Insulin Lispro | TI - B (1x30 U)/TI - A (2x15 U)/10 U sc Insulin Lispro
Started | 13 | 16
Completed | 13 | 14
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: TI Dosing Period 2 (1 Day)
Arm/Group | TI - A (2x15 U)/TI - B (1x30 U)/10 U sc Insulin Lispro | TI - B (1x30 U)/TI - A (2x15 U)/10 U sc Insulin Lispro
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0
Period: Washout 2 (3 - 14 Days)
Arm/Group | TI - A (2x15 U)/TI - B (1x30 U)/10 U sc Insulin Lispro | TI - B (1x30 U)/TI - A (2x15 U)/10 U sc Insulin Lispro
Started | 13 | 14
Completed | 12 | 14
Not Completed | 1 | 0
Not completed — Cannot Use Clamp Data | 1 | 0
Period: Lispro Dosing Period (1 Day)
Arm/Group | TI - A (2x15 U)/TI - B (1x30 U)/10 U sc Insulin Lispro | TI - B (1x30 U)/TI - A (2x15 U)/10 U sc Insulin Lispro
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Any subject that received at least one treatment with TI inhalation powder
Arm/Group | Safety Population
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m squared] | 26.61 (2.772)

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence of Two 15 U Cartridges (TI Inhalation Powder A) and One 30 U Cartridge (TI Inhalation Powder B) Based on Baseline Corrected Insulin AUC0-360
Description: Dose-normalized baseline-corrected area under the serum insulin vs. time curve
Time Frame: 0 to 360 minutes post-dose
Population: Per Protocol Population - All subjects who completed the crossover portion of the trial (through Visit 3), had serum insulin concentration data for both TI Inhalation Powder A and TI Inhalation Powder B and were deemed to be protocol compliant (no major protocol violations during the clinical trial).
Measure: Least Squares Mean (Standard Error); unit: (micro U)*min/mL
Groups:
- Techosphere Insulin - A (2 x 15 U): 30 U of Technosphere Insulin (TI) administered as 2 x 15 U cartridges as a single-dose during a glucose clamp procedure
- Techosphere Insulin - B (1 x 30 U): 30 U of Technosphere Insulin (TI) administered as 1 x 30 U cartridges as a single-dose during a glucose clamp procedure
Arm/Group | Techosphere Insulin - A (2 x 15 U) | Techosphere Insulin - B (1 x 30 U)
Number analyzed (Participants) | 25 | 25
(micro U)*min/mL | 3337.2 (1.096) | 3396.6 (1.096)
Statistical Analysis 1: Comparison: Techosphere Insulin - A (2 x 15 U) vs Techosphere Insulin - B (1 x 30 U); Test type: Superiority or Other; Ratio of Geometric Means = 0.982, 90% CI 2-sided [0.846 to 1.141] — Geometric Mean Ratio of serum insulin from a single 30 U cartridge to 2 x 15 U cartridges of TI. Based on pair-wise comparisons from analysis of covariance fitting the model: natural log of parameter = cohort, treatment, visit, subject (cohort)

2. Primary Outcome: Bioequivalence of Two 15 U Cartridges (TI Inhalation Powder A) and One 30 U Cartridge (TI Inhalation Powder B) Based on Baseline Corrected Insulin Cmax.
Description: Maximum observed baseline-corrected serum insulin concentration
Time Frame: 0 to 360 minutes post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: (micro U)/mL
Arm/Group | Techosphere Insulin - A (2 x 15 U) | Techosphere Insulin - B (1 x 30 U)
Number analyzed (Participants) | 25 | 25
(micro U)/mL | 65.72 (1.098) [0.823 to 1.099] | 69.08 (1.098)
Statistical Analysis 1: Comparison: Techosphere Insulin - A (2 x 15 U) vs Techosphere Insulin - B (1 x 30 U); Test type: Superiority or Other; Ratio of Geometric Means = 0.951, 90% CI 2-sided [0.823 to 1.099] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Bioequivalence of Two 15 U Cartridges (TI Inhalation Powder A) and One 30 U Cartridge (TI Inhalation Powder B) Based on Baseline Corrected Insulin Tmax
Time Frame: 0 to 360 minutes post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: min
Arm/Group | Techosphere Insulin - A (2 x 15 U) | Techosphere Insulin - B (1 x 30 U)
Number analyzed (Participants) | 25 | 25
min | 10 [5 to 24] | 10 [5 to 20]
Statistical Analysis 1: Comparison: Techosphere Insulin - A (2 x 15 U) vs Techosphere Insulin - B (1 x 30 U); Test type: Superiority or Other; p = 0.3531, Signed Rank Test; Median Difference (Final Values) = 0

4. Primary Outcome: Relative Bioavailability of 30 U of TI (TI Inhalation Powder B) Versus 10 U of sc Insulin Lispro
Description: Dose-normalized baseline-corrected area under the serum insulin vs. time curve (time 0 to 360 minutes post-dose)
Time Frame: 0 to 360 minutes post-dose
Population: Rapid-acting insulin Analogue (RAA) Population
  All subjects who had serum insulin concentration data for both TI Inhalation Powder B and insulin lispro and were deemed to be protocol compliant (no major protocol violations during the clinical trial).
Measure: Least Squares Mean (Standard Error); unit: (micro U)*min/mL
Groups:
- 10 U Subcutaneous (sc) Insulin Lispro: 10 U of insulin lispro administered subcutaneously during a glucose clamp procedure
Arm/Group | Techosphere Insulin - B (1 x 30 U) | 10 U Subcutaneous (sc) Insulin Lispro
Number analyzed (Participants) | 25 | 25
(micro U)*min/mL | 3406.8 (1.095) | 7404.0 (1.102)
Statistical Analysis 1: Comparison: Techosphere Insulin - B (1 x 30 U) vs 10 U Subcutaneous (sc) Insulin Lispro; Test type: Superiority or Other; Ratio of Geometric Means = 0.460, 90% CI 2-sided [0.366 to 0.578] — Geometric Mean Ratio of serum insulin from a single 30 U cartridge of TI to 10 U sc insulin lispro. Based on pair-wise comparisons from analysis of covariance fitting the model: natural log of parameter = cohort, treatment, visit, subject (cohort)

ADVERSE EVENTS:
Time Frame: From time of first dose to 30d after last dose; Serious adverse event (SAE) = until resolution
Arm/Group | Techosphere Insulin - A (2 x 15 U) | Techosphere Insulin - B (1 x 30 U) | 10 U Subcutaneous (sc) Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 9/27 | 14/29 | 5/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Techosphere Insulin - A (2 x 15 U) (N=27) | Techosphere Insulin - B (1 x 30 U) (N=29) | 10 U Subcutaneous (sc) Insulin Lispro (N=26)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0
Headache (Nervous system disorders) | 2 | 5 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.